CLINICAL TRIAL: NCT01099826
Title: Increasing CRC Screening in Primary Care Settings
Brief Title: Increasing Colorectal Cancer (CRC) Screening In Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: University of Illinois at Chicago (Other); Jesse Brown VA Medical Center (U.S. Federal Agency); University of Utah (Other); Vanderbilt University (Other); Penn State University (Other); Portland State University (Other)
Responsible Party: Principal Investigator, Usha Menon, Faculty, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: R01NR008425 (NIH)
Record Dates: First submitted 2010-04-06; First posted 2010-04-08 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Colorectal Cancer Screening
Keywords: colorectal cancer screening; tailored education; motivational interview; patient education
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- lifestyle counseling tailored (Experimental)
  Interventions: Behavioral: Tailored counseling
- lifestyle counseling motivational (Experimental)
  Interventions: Behavioral: Motivational Interview
- control (No Intervention)

INTERVENTIONS:
Behavioral: Tailored counseling — education tailored to baseline beliefs by trained counselor over phone
  Arms: lifestyle counseling tailored
Behavioral: Motivational Interview — motivational interview by trained MI counselors by phone
  Arms: lifestyle counseling motivational

SUMMARY:
Colorectal cancer screening remains lower than optimal. The purpose of this study was to test the efficacy of phone-based motivational interviewing versus tailored communication versus usual care in increasing CRC screening in primary care clinics.

DETAILED DESCRIPTION:
Regular screening reduces both morbidity and mortality from colorectal cancer (CRC). Screening rates, however, remain low suggesting the need for innovative research designed to increase screening behavior. The purpose of this study is to compare the effectiveness of two interventions (Tailored Health Communication [THC] and Motivational Interviewing [MI]) in increasing CRC screening behavior. Both interventions are based on a strong conceptual framework derived from the Health Belief Model (HBM) and Transtheoretical Model (TTM), allowing us to explore the underlying mechanisms through which these interventions impact behavior change.

The primary aim of this study is to compare CRC screening test use among 804 participants randomly allocated to control or intervention conditions; participants will be recruited from the two sites (Chicago, IL, and Nashville, TN). The 3 study groups will receive (1) standard care, (2) tailored health communication, and (3) motivational interviewing. Eligibility criteria for study participants includes being 50 years or older, not having CRC, and being of average or moderate risk for CRC. Study participants will be surveyed by telephone about CRC-related beliefs pre-intervention (Time 1), 1 month postintervention (Time 2), and at 6 months postintervention (Times 3 and 4, respectively). Dichotomous behavioral outcomes (had screening test or not) and stages of CRC screening test adoption (based on the TTM) will be assessed, as well as sociodemographic and belief predictors of screening behavior. Binomial and multinomial logistic regression models will be used to evaluate screening test use and stage of test adoption. Sociodemographic and belief variables will be used as covariates, with intervention group as the primary independent predictor. Descriptive statistics and ANOVA will be employed to assess between intervention differences in amenable beliefs. Path (mediation) analysis will be performed to further explore the underlying mechanisms through which THC and MI may differentially affect CRC screening behavior.

ELIGIBILITY:
Inclusion Criteria:

* all genders
* can speak, read, write English
* no diagnosis of colorectal cancer
* non-adherent with screening
* age 50 or older

Exclusion Criteria:

* had colorectal cancer
* adherent with screening

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2004-10; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
completing CRC screening test | 1 and 6 months post education

CONTACTS AND LOCATIONS:
Overall Officials: Usha Menon, PhD, Principal Investigator — Arizona State University

REFERENCES:
- [Background] Wahab S, Menon U, Szalacha L. Motivational interviewing and colorectal cancer screening: a peek from the inside out. Patient Educ Couns. 2008 Aug;72(2):210-7. doi: 10.1016/j.pec.2008.03.023. Epub 2008 May 8. PMID 18467066
- [Derived] Menon U, Belue R, Wahab S, Rugen K, Kinney AY, Maramaldi P, Wujcik D, Szalacha LA. A randomized trial comparing the effect of two phone-based interventions on colorectal cancer screening adherence. Ann Behav Med. 2011 Dec;42(3):294-303. doi: 10.1007/s12160-011-9291-z. PMID 21826576